CLINICAL TRIAL: NCT03000803
Title: Implications of Circadian Variation of Human Endocannabinoid Levels on Obesity Risk
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI is leaving the institution and study is being terminated with the IRB.
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB16-1174
Record Dates: First submitted 2016-12-12; First posted 2016-12-22 (Estimated); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Total Caloric Intake (Experimental): The Early Total Caloric Intake study group will consume the majority of their daily calories during breakfast.
  Interventions: Behavioral: Early Total Caloric Intake
- Late Total Caloric Intake (Active Comparator): The Late Total Caloric Intake study group will consume the majority of their daily calories during dinner.
  Interventions: Behavioral: Late Total Caloric Intake

INTERVENTIONS:
Behavioral: Early Total Caloric Intake — Provide subjects a regimented amount of calories at each meal.
  Arms: Early Total Caloric Intake
Behavioral: Late Total Caloric Intake — Provide subjects a regimented amount of calories at each meal.
  Arms: Late Total Caloric Intake

SUMMARY:
The purpose of this study is to examine how the timing of eating changes 24hr profiles of lipids involved in eating for pleasure and how the body makes and uses energy (metabolism).

DETAILED DESCRIPTION:
The timing of food intake and caloric distribution across the 24hr day are emerging as contributing factors to weight gain. The idea that not only what you eat, but when you eat can contribute to weight gain has garnered interest from both the scientific community and the public. In fact, the distribution of caloric intake over the 24hr day has been recently recognized as a potential source of "circadian misalignment" which can result in adverse health outcomes, including overeating, impaired glucose tolerance and insulin sensitivity. Moreover, reward driven eating (eating for the pleasurable aspect instead of energy need) generally results in caloric intake well in excess of energy requirements and is recognized as a major culprit in the epidemic of obesity. The endocannabinoid (eCB) system is involved in both homeostatic processes (energy need only) that govern food intake, and has been shown to play a key role in reward eating. Thus, the role of circadian organization of the eCB system and how misalignment may contribute to overeating, overweight, obesity, and diabetes is the main focus of this study. The overall goal is to determine whether the timing of food intake is a major determinant of the 24 hour variation in eCB activity that in turn affects hunger and appetite, glucose metabolism, and insulin sensitivity. This study will focus on overweight individuals who are at high risk of obesity but are still on a trajectory that can potentially be reversed by lifestyle changes. Following a careful assessment of the subject's habitual sleep and meal timing and caloric distribution under real life conditions, a short laboratory study will determine whether participants who consume more of their daily calories later in the day (later dietary chronotype) display delays in the eCB rhythm and lower insulin sensitivity. During a 6-day in patient intervention, combining laboratory and ambulatory procedures, study procedures will assess the effect of experimentally changing caloric distribution across the day, advancing versus delaying the dietary chronotype. The outcome measures will be the timing of the daily peak of the eCB rhythm and insulin sensitivity. Identification of circadian misalignment of the eCB system as a mediator of increased food intake and reduced insulin sensitivity may help develop novel preventive strategies.

ELIGIBILITY:
Inclusion Criteria:

* self-report sleeping between 7-hrs/night and 9-hrs/night, between 22:00 and 08:00
* no previously diagnosed sleep disorders (including obstructive sleep apnea (OSA))
* no existing diagnosis of prediabetes or diabetes
* no history of endocrine dysfunction
* no history of psychiatric, cardiovascular, or eating disorders
* must not have a gastro-intestinal disease that requires dietary adjustment
* currently taking no medications (including birth control)

Exclusion Criteria:

* drug and nicotine use, habitual alcohol use of more than 2 drinks per day, and caffeine intake of more than 300 mg per day
* anyone who has participated in medically managed weight loss program within the past year
* anyone who has undergone bariatric surgery
* must not have dietary restrictions
* must not work night shifts or crossed any time zones in the month prior to the study.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2026-10 (Estimated); Primary Completion 2029-10 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
Change in the time of acrophase of the 24hr eCB profile | Baseline to Day 38
  A shift in the timing ( time of day, h:mm) of the peak (acrophase) of the eCB rhythm.
Change in appetite/hunger and reward-related eating scores | Baseline to Day 38
  The change in the temporal profile of hunger and appetite ratings (measured at 6 time points over a 24hr period) as well as reward-related eating (RRE) from baseline to after the intervention. The ratings of hunger and appetite, and RRE from baseline to intervention will be measured by number rating, on a 10 point scale for hunger and appetite and agree/don't agree or a 5-point scale for the RREs.
Change in glucose tolerance | Baseline to Day 38
  The change in glucose tolerance from baseline to after the intervention will be measured. Glucose outcomes from CGM include Mean Absolute Glucose (MAG - mg/dl), Coefficient of Variation (CV - mg/dl), Standard Deviation (SD-mg/dl), Area Under the Curve (AUC - mg/dl), Time Spent in Range (TIR - minutes), Continuous Overall Net Glycemic Action (CONGA - (mg/dl) per minutes ).
Change in insulin sensitivity | Baseline to Day 38
  The change in insulin sensitivity from baseline to after the intervention will be measured. Insulin sensitivity measurements from the MMT include area under the curve for insulin (pmol/L) and cpeptide (pmol/L) as well as peak values (pmol/L).

SECONDARY OUTCOMES:
Change in Weight | Baseline to Day 38
  The change in weight (kilograms) from baseline after intervention will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Erin Hanlon, PhD, Principal Investigator — University of Chicago

IPD SHARING:
Plan to Share IPD: No
There is currently no plan to make IPD available to other researchers.